CLINICAL TRIAL: NCT02637687
Title: A Phase 1/2 Study of the Oral TRK Inhibitor Larotrectinib in Pediatric Patients With Advanced Solid or Primary Central Nervous System Tumors
Brief Title: A Study to Test the Safety and Efficacy of the Drug Larotrectinib for the Treatment of Tumors With NTRK-fusion in Children
Acronym: SCOUT
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20290; LOXO-TRK-15003 (Other: Loxo Oncology, Inc); 2022-502668-20-00 (Other: CTIS (EU)); 2016-003498-16 (EudraCT Number)
Record Dates: First submitted 2015-12-10; First posted 2015-12-22 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors Harboring NTRK Fusion
Keywords: Advanced solid tumors; Central nervous system (CNS) tumor; Extra-cranial tumor; Infantile fibrosarcoma (IFS); Neurotrophic tyrosine receptor kinase (NTRK); NTRK1; NTRK2; NTRK3; Fusion Positive; TRK fusion; TRKA; TRKB; TRKC; ETV6
MeSH Terms: conditions — Neoplasms | interventions — larotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (6):
- Phase 1 dose escalation (Experimental): Patients will receive the different levels of dose on Day 1 (BID in accordance with the cohort assignment). Each cycle will consist of 28 days of continuous dosing.
  Individual patients will continue daily larotrectinib dosing until PD, unacceptable toxicity, or other reason for treatment discontinuation. (arm closed)
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Phase 1 dose expansion (Experimental): Patients who are enrolled in the expansion cohort, following the formal dose escalation phase of the study.
  Distinct from the Phase 1 dose escalation cohort, the Phase 1 expansion cohort will enroll pediatric patients with advanced solid or primary CNS tumors with a documented NTRK gene fusion, or in the case of IFS, CMN or SBC with documented ETV6 rearrangement by FISH or RT-PCR or a documented NTRK fusion by NGS.
  This expansion cohort will follow the same schedule of assessments as the dose escalation cohorts. (arm closed)
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Phase 2: Patients with tumors bearing NTRK fusions (IFS)_Cohort 1 (Experimental): Patients will receive larotrectinib dose on Day 1 (BID in accordance with the cohort assignment) at the recommended Phase 2 dose as determined in the Phase 1 portion of this study. Each cycle will consist of 28 days of continuous dosing.
  Individual patients will continue daily larotrectinib dosing until PD, unacceptable toxicity, or other reason for treatment discontinuation. (arm closed)
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Phase 2: Other extra-cranial solid tumors_Cohort 2 (Experimental): Patients will receive larotrectinib dose on Day 1 (BID in accordance with the cohort assignment) at the recommended Phase 2 dose as determined in the Phase 1 portion of this study. Each cycle will consist of 28 days of continuous dosing.
  Individual patients will continue daily larotrectinib dosing until PD, unacceptable toxicity, or other reason for treatment discontinuation. (arm closed)
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Phase 2: Primary CNS tumors_Cohort 3 (Experimental): Patients will receive larotrectinib dose on Day 1 (BID in accordance with the cohort assignment) at the recommended Phase 2 dose as determined in the Phase 1 portion of this study. Each cycle will consist of 28 days of continuous dosing.
  Individual patients will continue daily larotrectinib dosing until PD, unacceptable toxicity, or other reason for treatment discontinuation.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Phase 2: Bone health assessment_sub-cohort (Experimental): Patients will receive larotrectinib dose on Day 1 (BID in accordance with the cohort assignment) at the recommended Phase 2 dose as determined in the Phase 1 portion of this study. Each cycle will consist of 28 days of continuous dosing.
  Individual patients will continue daily larotrectinib dosing until PD, unacceptable toxicity, or other reason for treatment discontinuation.
  Patients in this group will undergo bone health assessments in addition to all other efficacy and safety assessments.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)

INTERVENTIONS:
Drug: Larotrectinib (Vitrakvi, BAY2757556) — BAY2757556 will be administered orally as capsule or in liquid form over continuous 28-day cycles.
  Other Names: LOXO-101

SUMMARY:
The study is being done to test the safety of a cancer drug called larotrectinib in children. The cancer must have a change in a particular gene (NTRK1, NTRK2 or NTRK3). Larotrectinib blocks the actions of these NTRK genes in cancer cells and can therefore be used to treat cancer.

The first study part (Phase 1) is done to determine what dose level of larotrectinib is safe for children, how the drug is absorbed and changed by their bodies and how well the cancer responds to the drug. The main purpose of the second study part (Phase 2) is to investigate how well and how long different cancer types respond to the treatment with larotrectininb.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 (Closed):

  * Dose escalation: Birth through 21 years of age at C1D1 with a locally advanced or metastatic solid tumor or primary CNS tumor that has relapsed, progressed or was nonresponsive to available therapies and for which no standard or available systemic curative therapy exists; OR Infants from birth and older with a diagnosis of malignancy and with a documented NTRK fusion that has progressed or was nonresponsive to available therapies, and for which no standard or available curative therapy exists; OR Patients with locally advanced infantile fibrosarcoma who would require, in the opinion of the investigator, disfiguring surgery or limb amputation to achieve a complete surgical resection. Phase I dose escalation cohorts are closed to enrollment.
  * Dose expansion: In addition to the above stated inclusion criteria, patients must have a malignancy with a documented NTRK gene fusion with the exception of patients with infantile fibrosarcoma, congenital mesoblastic nephroma or secretory breast cancer. Patients with infantile fibrosarcoma, congenital mesoblastic nephroma or secretory breast cancer may enroll into this cohort with documentation of an ETV6 rearrangement by FISH or RT-PCR or a documented NTRK fusion by next generation sequencing.
* Phase 2:

  -- Infants from birth and older at C1D1 with a locally advanced or metastatic infantile fibrosarcoma, patients with locally advanced infantile fibrosarcoma who would require, in the opinion of the investigator, disfiguring surgery or limb amputation to achieve a complete surgical resection; OR Birth through 21 years of age at C1D1 with a locally advanced or metastatic solid tumor or primary CNS tumor that has relapsed, progressed or was nonresponsive to available therapies and for which no standard or available systemic curative therapy exists with a documented NTRK gene fusion (or in the case of infantile fibrosarcoma, congenital mesoblastic nephroma or secretory breast cancer with documented ETV6 rearrangement (or NTRK3 rearrangement after discussion with the sponsor) by FISH or RT-PCR. Patients with NTRK-fusion positive benign tumors are also eligible; OR Potential patients older than 21 years of age with a tumor diagnosis with histology typical of a pediatric patient and an NTRK fusion may be considered for enrollment following discussion between the local site Investigator and the Sponsor.
* Patients with primary CNS tumors or cerebral metastasis
* Karnofsky (those 16 years and older) or Lansky (those younger than 16 years) performance score of at least 50.
* Adequate hematologic function
* Adequate hepatic and renal function

Exclusion Criteria:

* Major surgery within 14 days (2 weeks) prior to C1D1
* Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to C1D1, ongoing cardiomyopathy; current prolonged QTc interval > 480 milliseconds
* Active uncontrolled systemic bacterial, viral, or fungal infection
* Current treatment with a strong CYP3A4 inhibitor or inducer. Enzyme-inducing anti-epileptic drugs (EIAEDs) and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed.
* Phase 2 only:

  * Prior progression while receiving approved or investigational tyrosine kinase inhibitors targeting TRK, including entrectinib, crizotinib and lestaurtinib. Patients who received a TRK inhibitor for less than 28 days of treatment and discontinued because of intolerance remain eligible.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of participants in an assigned dose cohort with treatment emergent adverse events (TEAEs) by grade assessed by NCI-CTCAE v 4.03 who experience a DLT | From Day 1 to Day 28 of Cycle 1 (1 Cycle=28 days)
  DLT: Dose-limiting toxicity. NCI-CTCAE: National Cancer Institute-Common Terminology Criteria for Adverse Events.
Phase 1: Number of participants with TEAEs | From first dose of larotrectinib up to 93 months
Phase 1: Severity of TEAEs | From first dose of larotrectinib up to 93 months
Phase 2: Overall response rate (ORR) by IRRC | From first dose of Larotrectinib to disease progression or subsequent therapy or surgical intervention or death, up to 76 months
  Proportion of participants with a best overall response of complete response (CR) or partial response (PR) as determined by an independent radiology review committee (IRRC) based on Response Evaluation Criteria in Solid Tumours (RECIST) 1.1, Response Assessment in Neuro Oncology (RANO) or International Neuroblastoma Response Criteria (INRC) as appropriate to tumor type who express NTRK gene fusions.

SECONDARY OUTCOMES:
Phase 1: Maximum concentration of larotrectinib in plasma (Cmax) | Cohort 1 and 2: Cycle 1 Day 1 (C1D1) at 1 and 4 hours post-dose and C2D1 at pre-dose, and at 1 and 4 hours post-dose; Cohort 3 and Dose Expansion Cohort: C1D1 at 1 and 4 hours post-dose and C4D1 at pre-dose, 1 and 4 hours post-dose
Phase 1: Area under the concentration versus time curve from time 0 to t (AUC0-t) of larotrectinib in plasma | Cohort 1 and 2: C1D1 at 1 and 4 hours post-dose and C2D1 at pre-dose, and at 1 and 4 hours post-dose; Cohort 3 and Dose Expansion Cohort: C1D1 at 1 and 4 hours post-dose and C4D1 at pre-dose, 1 and 4 hours post-dose
Phase 1: Oral clearance (CL/F) | Cohort 1 and 2: C1D1 at 1 and 4 hours post-dose and C2D1 at pre-dose, and at 1 and 4 hours post-dose; Cohort 3 and Dose Expansion Cohort: C1D1 at 1 and 4 hours post-dose and C4D1 at pre-dose, 1 and 4 hours post-dos
Phase 1: Cerebral spinal fluid/plasma ratio of larotrectinib | C1D1 in conjunction with the post-dose 1-hour PK sample
Phase 1: Maximum tolerated dose (MTD) | From C1D1 to C1D28 of treatment of each participant in each of the assigned dose cohort, up to 16 months
Phase 1: Recommended dose for Phase 2 | From the date a participants from assigned Cohort was administered the first dose to the date of the last dose for the last patient from the dose escalation phase, up to 16 months
Phase 1: Overall Response Rate (ORR) | From first dose of Larotrectinib to disease progression or subsequent therapy or surgical intervention or death (due to any cause), up to 93 months
  Proportion of participants with best overall response (BOR) of CR and PR; PFS, CBR and maximum change in tumor burden as assessed based on RECIST 1.1, INRC or RANO as appropriate for tumor type by IRRC.
Phase 1: Mean change from baseline in Pain scores as assessed by the Wong-Baker Faces scale | Baseline and D1 of every cycle (1 Cycle=28 days), up to 93 months
  Wong-Baker Faces Scale giving a pain scale between 0 (no hurt) to 10 (hurts worst).
Phase 1: Mean change in Health-related quality of life scores by PedsQL-Core | Baseline and D1 of every cycle (1 Cycle=28 days), Up to 93 months
  The health-related quality of life (HRQoL) is assessed with the Pediatrics Quality of Life - Core Module (PedsQL-Core) questionnaire that consists of various age-related items regarding physical, emotional, social and school functioning and gives an overall score between 0 (highest HRQoL) and 144 (lowest HRQoL).
Phase 2: Best overall response (BOR) | From first dose of Larotrectinib to disease progression or subsequent therapy or surgical intervention or death (due to any cause), up to 76 months
  Participants with best overall response (BOR) of either CR or PR determined by Investigator's or IRC's response assessment based on RANO, INRC and RECIST 1.1 as appropriate for tumor type
Phase 2: Duration of response (DOR) | From start of first objective response of confirmed CR or PR to progression or death (due to any cause), up to 76 months
  DOR determined by 1) an independent radiology review committee and 2) the treating Investigator.
Phase 2: Proportion of patients with any tumor regression (i.e., any decrease from baseline of the longest diameters of target lesions) as a best response | From first dose of Larotrectinib, up to 76 months
Phase 2: Progression-free survival (PFS) | From first dose of Larotrectinib to disease progression or subsequent therapy or surgical intervention or death (due to any cause), up to 112 months
Phase 2: Overall survival (OS) | From first dose of Larotrectinib to death (due to any cause), up to 112 months
Phase 2: Number of participants with Treatment emergent adverse events (TEAEs) | From first dose of larotrectinib to discontinuation of treatment or death (due to any cayse), up to 112 months
Phase 2: Severity of adverse events as assessed by NCI-CTCAE grading V 4.03 | From first dose of larotrectinib to discontinuation of treatment or death (due to any cause), up to 112 months
Phase 2: Clinical Benefit Rate (CBR) | From first dose of Larotrectinib to disease progression or subsequent therapy or surgical intervention or death (due to any cause), up to 76 months
  CBR (i.e., best overall response of CR, PR or SD lasting 16 weeks or more as determined by 1) an independent radiology review committee (IRC) and 2) by the treating Investigator.
Phase 2: Concordance coefficient | From baseline/screening and if feasible end of treatment (EOT) and or PD and or at re-start of study treatment following a "drug holiday" and disease recurrence, up to 112 months
  Concordance coefficient of intra-patient molecular profile
Phase 2: Post-operative tumor staging | From first dose of Larotrectinib to surgical intervention, up to 112 months
  Post-operative stage in patients treated with larotrectinib according to the TNM Classification of malignant tumors of the Union for International Cancer Control (UICC).
Phase 2: Post-operative surgical margin assessment | From first dose of Larotrectinib to surgical intervention, up to 112 months
  Surgical margin status in patients treated with larotrectinib using the International Cancer Control (UICC)-R classification and the Intergroup Rhabdomyosarcoma Staging (IRS) systems.
Phase 2: Pre-treatment surgical plan to preserve function and cosmetic outcome | From first dose of Larotrectinib to surgical intervention, up to 112 months
  Descriptive analysis of pretreatment surgical plan.
Phase 2: Post-treatment plans to conserve function and cosmetic outcome | From surgical intervention to subsequent therapy, up to 112 months
  Descriptive analysis of post-treatment plans

CONTACTS AND LOCATIONS:
Locations (45):
- United States (11):
  - Children's Hospital Los Angeles - Hematology/Oncology, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Lucille Packard Children's Hospital Stanford - Pediatric Nephrology, Palo Alto, California
  - Nemours Children's Hospital - Florida - Hematology / Oncology, Orlando, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center New York - Main Campus, New York, New York
  - Cincinnati Children's Hospital Medical Center | Division of Nephrology and Hypertension, Cincinnati, Ohio
  - Children's Hospital of Philadelphia - Hematology/Oncology, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hosptial - Oncology, Seattle, Washington
- Australia (3):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital Melbourne, Parkville, Victoria
- Canada (3):
  - BC Children's Hospital - Hematology/Oncology, Vancouver, British Columbia
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- China (3):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
- Czechia (2):
  - FN Brno - Detska nemocnice, Brno
  - Fakultni nemocnice v Motole, Prague
- Rigshospitalet - Børn og Unge, Copenhagen, Denmark
- France (2):
  - Institut Curie - Ulm - Paris, Paris
  - Gustave Roussy - Departement Oncologie-Radiotherapie, Villejuif
- Germany (3):
  - Universitaetsklinikum Heidelberg - KiTZ | Klinik für Paediatrische Onkologie, Haematologie, Immunologie und Pneumologie, Heidelberg, Baden-Wurttemberg
  - KLINIKUM STUTTGART - Olgahospital | Paediatrie 5 (Onkologie, Haematologie, Immunologie), Stuttgart, Baden-Wurttemberg
  - Charité - Campus Virchow-Klinikum (CVK), Klinik für Pädiatrie mit Schwerpunkt Onkologie und Hämatologie, Berlin
- Children's Health Ireland Crumlin, Crumlin, Dublin, Ireland
- Clalit Health Services Schneider Children's Medical Center, Petah Tikva, Israel
- Fondazione IRCCS Istituto Nazionale dei Tumori - S. C. Pediatria Oncologica, Milan, Lombardy, Italy
- Japan (3):
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
- Prinses Maxima Centrum, Utrecht, Netherlands
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona, Spain
- Karolinska Universitetssjukhuset i Solna, Stockholm, Sweden
- Universitätskinderspital Zürich, Zurich, Switzerland
- Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul, Turkey (Türkiye)
- Ukraine (2):
  - Governmental Noncommercial Institution "National Cancer Institute, Kyiv
  - Western Ukrainian Specialized Pediatric Medial Centre, Surgical Department, Lviv
- Royal Marsden NHS Trust (Surrey), Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Brose MS, Westphalen CB, Pan X, Bernard-Gauthier V, Kurtinecz M, Guo H, Aris V, Brett NR, Majdi A, Subbiah V, Pennell NA, Kehl KL, Drilon A. Larotrectinib Compared With Real-World Non-Tropomyosin Receptor Kinase Inhibitor Therapies in Patients With Tropomyosin Receptor Kinase Fusion Cancer. JCO Precis Oncol. 2025 Apr;9:e2400500. doi: 10.1200/PO-24-00500. Epub 2025 Apr 23. PMID 40267388
- [Derived] Mascarenhas L, DuBois SG, Albert CM, Bielack S, Orbach D, Federman N, Geoerger B, Nagasubramanian R, Zhang Y, Chisholm J, Gallego Melcon S, Goto H, Morgenstern DA, Owens C, Pappo AS, Perreault S, Schulte JH, Shukla N, Zwaan CM, Neu N, Bernard-Gauthier V, De La Cuesta E, van Tilburg CM, Laetsch TW. Elective Discontinuation of Larotrectinib in Pediatric Patients With TRK Fusion Sarcomas and Related Mesenchymal Tumors. J Clin Oncol. 2025 Apr;43(10):1180-1187. doi: 10.1200/JCO.24.00848. Epub 2025 Jan 27. PMID 39869835
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] Kummar S, Shen L, Hong DS, McDermott R, Keedy VL, Casanova M, Demetri GD, Dowlati A, Melcon SG, Lassen UN, Leyvraz S, Liu T, Moreno V, Patel J, Patil T, Mallick AB, Sousa N, Tahara M, Ziegler DS, Norenberg R, Arvis P, Brega N, Drilon A, Tan DSW. Larotrectinib efficacy and safety in adult patients with tropomyosin receptor kinase fusion sarcomas. Cancer. 2023 Dec 1;129(23):3772-3782. doi: 10.1002/cncr.35036. Epub 2023 Sep 28. PMID 37769113
- [Derived] Bokemeyer C, Paracha N, Lassen U, Italiano A, Sullivan SD, Marian M, Brega N, Garcia-Foncillas J. Survival Outcomes of Patients With Tropomyosin Receptor Kinase Fusion-Positive Cancer Receiving Larotrectinib Versus Standard of Care: A Matching-Adjusted Indirect Comparison Using Real-World Data. JCO Precis Oncol. 2023 Jan;7:e2200436. doi: 10.1200/PO.22.00436. PMID 36689698
- [Derived] Rudzinski ER, Drilon A, Moore A, Spinosa S, Willi M, Laetsch TW. Testing methods to diagnose TRK fusion cancer - a plain language summary and patient perspective. Future Oncol. 2022 Dec;18(38):4141-4151. doi: 10.2217/fon-2022-0863. Epub 2023 Jan 6. PMID 36606522
- [Derived] Doz F, van Tilburg CM, Geoerger B, Hojgaard M, Ora I, Boni V, Capra M, Chisholm J, Chung HC, DuBois SG, Gallego-Melcon S, Gerber NU, Goto H, Grilley-Olson JE, Hansford JR, Hong DS, Italiano A, Kang HJ, Nysom K, Thorwarth A, Stefanowicz J, Tahara M, Ziegler DS, Gavrilovic IT, Norenberg R, Dima L, De La Cuesta E, Laetsch TW, Drilon A, Perreault S. Efficacy and safety of larotrectinib in TRK fusion-positive primary central nervous system tumors. Neuro Oncol. 2022 Jun 1;24(6):997-1007. doi: 10.1093/neuonc/noab274. PMID 34850167
- [Derived] Bebb DG, Banerji S, Blais N, Desmeules P, Gill S, Grin A, Feilotter H, Hansen AR, Hyrcza M, Krzyzanowska M, Melosky B, Noujaim J, Purgina B, Ruether D, Simmons CE, Soulieres D, Torlakovic EE, Tsao MS. Canadian Consensus for Biomarker Testing and Treatment of TRK Fusion Cancer in Adults. Curr Oncol. 2021 Jan 15;28(1):523-548. doi: 10.3390/curroncol28010053. PMID 33467570
- [Derived] Perreault S, Chami R, Deyell RJ, El Demellawy D, Ellezam B, Jabado N, Morgenstern DA, Narendran A, Sorensen PHB, Wasserman JD, Yip S. Canadian Consensus for Biomarker Testing and Treatment of TRK Fusion Cancer in Pediatric Patients. Curr Oncol. 2021 Jan 9;28(1):346-366. doi: 10.3390/curroncol28010038. PMID 33435412
- [Derived] Bielack SS, Cox MC, Nathrath M, Apel K, Blattmann C, Holl T, Jenewein R, Klenk U, Klothaki P, Muller-Abt P, Ortega-Lawerenz S, Reynolds M, Scheer M, Simon-Klingenstein K, Stegmaier S, Tupper R, Vokuhl C, von Kalle T. Rapid, complete and sustained tumour response to the TRK inhibitor larotrectinib in an infant with recurrent, chemotherapy-refractory infantile fibrosarcoma carrying the characteristic ETV6-NTRK3 gene fusion. Ann Oncol. 2019 Nov;30 Suppl 8:viii31-viii35. doi: 10.1093/annonc/mdz382. Epub 2019 Dec 24. PMID 32223937
- [Derived] Hong DS, DuBois SG, Kummar S, Farago AF, Albert CM, Rohrberg KS, van Tilburg CM, Nagasubramanian R, Berlin JD, Federman N, Mascarenhas L, Geoerger B, Dowlati A, Pappo AS, Bielack S, Doz F, McDermott R, Patel JD, Schilder RJ, Tahara M, Pfister SM, Witt O, Ladanyi M, Rudzinski ER, Nanda S, Childs BH, Laetsch TW, Hyman DM, Drilon A. Larotrectinib in patients with TRK fusion-positive solid tumours: a pooled analysis of three phase 1/2 clinical trials. Lancet Oncol. 2020 Apr;21(4):531-540. doi: 10.1016/S1470-2045(19)30856-3. Epub 2020 Feb 24. PMID 32105622
- [Derived] Bielack SS, Cox MC, Nathrath M, Apel K, Blattmann C, Holl T, Jenewein R, Klenk U, Klothaki P, Muller-Abt P, Ortega-Lawerenz S, Reynolds M, Scheer M, Simon-Klingenstein K, Stegmaier S, Tupper R, Vokuhl C, von Kalle T. Rapid, complete and sustained tumour response to the TRK inhibitor larotrectinib in an infant with recurrent, chemotherapy-refractory infantile fibrosarcoma carrying the characteristic ETV6-NTRK3 gene fusion. Ann Oncol. 2019 Nov 1;30(Suppl_8):viii31-viii35. doi: 10.1093/annonc/mdz382. PMID 31738425
- [Derived] DuBois SG, Laetsch TW, Federman N, Turpin BK, Albert CM, Nagasubramanian R, Anderson ME, Davis JL, Qamoos HE, Reynolds ME, Cruickshank S, Cox MC, Hawkins DS, Mascarenhas L, Pappo AS. The use of neoadjuvant larotrectinib in the management of children with locally advanced TRK fusion sarcomas. Cancer. 2018 Nov 1;124(21):4241-4247. doi: 10.1002/cncr.31701. Epub 2018 Sep 11. PMID 30204247
- [Derived] Laetsch TW, DuBois SG, Mascarenhas L, Turpin B, Federman N, Albert CM, Nagasubramanian R, Davis JL, Rudzinski E, Feraco AM, Tuch BB, Ebata KT, Reynolds M, Smith S, Cruickshank S, Cox MC, Pappo AS, Hawkins DS. Larotrectinib for paediatric solid tumours harbouring NTRK gene fusions: phase 1 results from a multicentre, open-label, phase 1/2 study. Lancet Oncol. 2018 May;19(5):705-714. doi: 10.1016/S1470-2045(18)30119-0. Epub 2018 Mar 29. PMID 29606586
- [Derived] Drilon A, Laetsch TW, Kummar S, DuBois SG, Lassen UN, Demetri GD, Nathenson M, Doebele RC, Farago AF, Pappo AS, Turpin B, Dowlati A, Brose MS, Mascarenhas L, Federman N, Berlin J, El-Deiry WS, Baik C, Deeken J, Boni V, Nagasubramanian R, Taylor M, Rudzinski ER, Meric-Bernstam F, Sohal DPS, Ma PC, Raez LE, Hechtman JF, Benayed R, Ladanyi M, Tuch BB, Ebata K, Cruickshank S, Ku NC, Cox MC, Hawkins DS, Hong DS, Hyman DM. Efficacy of Larotrectinib in TRK Fusion-Positive Cancers in Adults and Children. N Engl J Med. 2018 Feb 22;378(8):731-739. doi: 10.1056/NEJMoa1714448. PMID 29466156